CLINICAL TRIAL: NCT03381638
Title: Understanding Concussion/Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Blinktbi, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1415-14d
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Traumatic Brain Injury; Concussion, Brain
Keywords: Concussion; TBI; Sports; Medical Device; Fast
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Volunteer: Volunteers who report to have never had a concussion and are not at high risk of getting a concussion are scanned to obtain a baseline of all ages, sex, race, etc. All patients will be scanned with the Blink Reflexometer.
  Interventions: Device: Blink Reflexometer
- Concussion Protocol: Athletes who had a potential concussion and will go through any stage of the approved protocol, are scanned by the Blink Reflexometer device. Results are then analyzed prior to unblinding the clinical diagnosis from an Athletic Trainer and/or Neurologist.
  Interventions: Device: Blink Reflexometer

INTERVENTIONS:
Device: Blink Reflexometer — The device uses 5 light puffs of air to the side of the eye causing a blink reflex that is captured by the high-speed camera tracking the eyelids.

SUMMARY:
Using the Blink Reflexometer, athletes are scanned if they are potentially thought to have a concussion during a game or practice.

DETAILED DESCRIPTION:
In a blinded trial, any patient who during a game or practice situation had head contact, thus possible Traumatic Brain Injury (TBI) aka Concussion, in addition to the current approved protocols, patients are scanned with the Blink Reflexometer. Results are not available until the end of the season, thus eliminating the potential of someone relying on the results. The Blink Reflexometer uses 5 puffs of air on the side of the eye over 20 seconds. The air causes a blink reflex which is being correlated to a concussion. The results of the blink post concussion are compared to a baseline scan taken at the beginning of the season.

ELIGIBILITY:
Inclusion Criteria:

* Read, understand and sign patient consent (parent approval needed when pt is under 18yo)

Exclusion Criteria:

* Diagnosed concussion in past 4 weeks
* Ingesting any drugs banned by the US Anti-doping Association (USADA)
* Never prior diagnosed with a neurological abnormality, including Alzheimer's, MS, Huntington's, Epilepsy, etc.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers with a minimum age of 14yo. Any sex, nationality, sport played, etc are accepted.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Accuracy of Concussion Diagnosis | Data unblinded May 1, 2018 or at completion of season, which ever comes first.
  The results from the Blink machine should match the physicians diagnosis.

SECONDARY OUTCOMES:
Contributing Factors | Data unblinded May 1, 2018 or at completion of season, which ever comes first.
  There are a number of factors that could possible change the blink reflex such as Caffeine and Tobacco. We are capturing this data to confirm that the device can be accurate despite a patient ingesting these items.
Average Baseline | Data unblinded May 1, 2018 or at completion of season, which ever comes first.
  The goal is to eliminate the need for requiring a baseline scan on a patient in order to decide if they have a concussion or not. By scanning a large number of normal volunteers at various ages, sex, race, etc, we expect to see trends based on these factors.

CONTACTS AND LOCATIONS:
Overall Officials: Dena Garner, Ph.D., Principal Investigator — The Citadel
Locations (5):
- United States (5):
  - Johnson. C. Smith University, Charlotte, North Carolina
  - Hershey Bears Ice Hockey Team, Hershey, Pennsylvania
  - The Citadel, Charleston, South Carolina
  - South Carolina Stingrays, North Charleston, South Carolina
  - Spartinburg High School, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
All patient data will be anonymized prior to dissemination. Contact the sponsor for further details.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and ICF are available any time.
Access Criteria: Case by case basis.
URL: http://www.blinktbi.com

REFERENCES:
- [Background] Tsai NT, Goodwin JS, Semler ME, Kothera RT, Van Horn M, Wolf BJ, Garner DP. Development of a Non-Invasive Blink Reflexometer. IEEE J Transl Eng Health Med. 2017 Dec 19;5:3800204. doi: 10.1109/JTEHM.2017.2782669. eCollection 2017. PMID 29285420
- [Result] Garner, Goodwin, Tsai et al., Blink reflex parameters in baseline, active, and head-impact Division I athletes, Cogent Engineering, 2018; 5; 1429110